CLINICAL TRIAL: NCT06235944
Title: The Efficacy of Post-operative Analgesia of Sacral Erector Spinae Plane Block Versus Caudal Block in Penile Surgeries in Pediatrics
Brief Title: Sacral Erector Spinae Plane Block Versus Caudal Block in Penile Surgeries in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Allah Hamdy Elbahy, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 34989/10/21
Record Dates: First submitted 2024-01-22; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Sacral Erector Spinae Plane Block; Caudal Block; Penile Surgeries; Pediatrics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal block (Experimental): Patients were received (plain bupivacaine 0.25% 1 mg/kg + 2 % lidocaine 3 mg /kg) in total volume 1ml/ kg max 20 ml via Ultrasound Guided caudal Block.
  Interventions: Procedure: Caudal block
- Sacral erector spinae (Experimental): Patients were received (plain bupivacaine 0.25% 1 mg/kg + 2 % lidocaine 3 mg /kg) in total volume of 1 ml/ kg maximum 20ml divided in both sides via ultrasound guided sacral erector spinae plain block (ESPB).
  Interventions: Procedure: Sacral erector spinae block

INTERVENTIONS:
Procedure: Caudal block — Patients were received (plain bupivacaine 0.25% 1 mg/kg + 2 % lidocaine 3 mg /kg) in total volume 1ml/ kg max 20 ml via Ultrasound Guided caudal Block.
  Arms: Caudal block
Procedure: Sacral erector spinae block — Patients were received (plain bupivacaine 0.25% 1 mg/kg + 2 % lidocaine 3 mg /kg) in total volume of 1 ml/ kg maximum 20ml divided in both sides via ultrasound guided sacral erector spinae plain block (ESPB).
  Arms: Sacral erector spinae

SUMMARY:
The study will be conducted to compare the efficacy of ultrasound guided Sacral Erector Spinae Plane Block to caudal block on pain management in penile surgeries in pediatrics.

DETAILED DESCRIPTION:
The erector spinae plane block (ESPB) is a relatively new interfacial plane block that is used for postoperative analgesia in penile surgeries in pediatrics.

The sacral ESPB is a technique known to block the posterior branches of the sacral nerves. Also it blocks the lumbosacral plexus especially the sacral spinal nerves (S2_S4) when applied to high levels.

Caudal epidural block in children is one of the most widely administrated technique of regional anesthesia; it is an efficient way to offer perioperative analgesia for painful sub umbilical interventions. It enables early ambulation, hemodynamic stability and spontaneous breathing in patient groups at maximum risk of difficult airway.

Caudal block is a known worldwide technique but with some risks such as subdural, intra vascular injection, infection, injury to the nerve root or local anesthesia. Therefore, we try a new technique as sacral ESPB.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3 to 6 years.
* Male children.
* American Society of Anesthesiologists (ASA) I - II.
* Male who admitted for penile surgeries.

Exclusion Criteria:

* Parents who refused regional anesthesia.
* Patients presented with symptoms or signs of increased intracranial tension.
* Patients presented with advanced kidney, cardiac or liver diseases.
* Coagulation and bleeding disorders.
* Patients presented with skin or soft tissue infection at the proposed site of needle Insertion.
* Pre-existing neurologic disease (e.g. lower extremity peripheral neuropathy).
* Patients with known allergy to study drugs.
* Patints with developmental or mental delay.

Ages: 3 Years to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male children who undergoing penile surgery.
Enrollment: 70 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesic. | 24 hours postoperatively
  The time to first rescue analgesia was measured from the end to surgery till first dose of paracetamol administrated.

SECONDARY OUTCOMES:
Total rescue analgesia consumption | 24 hours postoperatively
  Total analgesic consumption (postoperative paracetamol IV 15 mg/kg) used if FLACC was 4 or more.
  The Face, Legs, Activity, Cry and Consolability (FLACC) scale is an observational scale The range from 0 to 10 with 0 representing no pain, 10 representing the worst pain
The degree of pain | 24 hours postoperatively
  The degree of pain was assessed after surgery over 24 hours using Face, Legs, Activity, Cry and Consolability (FLACC) score at time (30 minutes postoperative, 2, 4, 6, 12, 18, 24 hours).
  FLACC score is used for pain assessment in children between age of 3 to 6 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0 to 10 with 0 representing no pain, 10 representing the worst pain and we start to give rescue analgesia at score 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author